CLINICAL TRIAL: NCT01099670
Title: A Double-blind, Placebo-controlled, Randomised, Parallel-group, Dose-escalating, Repeat Dose Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacodynamic Effects and Pharmacokinetics of the Once Daily Rectal Application of 7.5, 10, 12.5 or 15 mg NRL001 in a 2 g Suppository for 14 Days
Brief Title: Safety, Tolerability, Pharmacodynamic and Pharmacokinetics of 7.5, 10, 12.5 or 15 mg NRL001 in a 2 g Suppository for 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRL001-01/2009 (SURD); 2009-017473-37 (EudraCT Number)
Record Dates: First submitted 2010-02-15; First posted 2010-04-07 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 7.5 mg NRL001 (Experimental): Nine subjects will receive 7.5 mg NRL001 in a 2 g suppository; three will receive matching placebo.
  Interventions: Drug: NRL001; Drug: Placebo
- 10 mg NRL001 (Experimental): Nine subjects will receive 10 mg NRL001 in a 2 g suppository; three will receive matching placebo.
  Interventions: Drug: NRL001; Drug: Placebo
- 12.5 mg NRL001 (Experimental): Nine subjects will receive 12.5 mg NRL001 in a 2 g suppository; three will receive matching placebo.
  Interventions: Drug: NRL001; Drug: Placebo
- 15 mg NRL001 (Experimental): Nine subjects will receive 15 mg NRL001 in a 2 g suppository; three will receive matching placebo.
  Interventions: Drug: NRL001; Drug: Placebo

INTERVENTIONS:
Drug: NRL001 — Rectal suppository Placebo
Drug: Placebo — Placebo

SUMMARY:
Healthy subjects will receive NRL001 or placebo once daily for 14 days. The four treatment groups, shown below, will each consist of 12 subjects:

Group 1; Nine subjects will receive a dose of 7.5 mg NRL001 in a 2 g suppository and three will receive matching placebo.

Group 2; Nine subjects will receive a dose of 10 mg NRL001 in a 2 g suppository and three will receive matching placebo.

Group 3; Nine subjects will receive a daily dose of 12.5 mg NRL001 in a 2 g suppository and three will receive matching placebo.

Group 4; Nine subjects will receive a daily dose of 15 mg NRL001 in a 2 g suppository and three will receive matching placebo.

The dosing of each group will be completed prior to the next group being dosed. Dose escalation will be dependent on a positive assessment of the safety profile of the preceding group by the Safety Monitoring Board.

The pharmacokinetics of NRL001 will be determined on Days 1, 7 and 14. Pharmacodynamics will be examined using a three lead Holter monitor at screening and at intervals throughout the study period. Adverse events, vital signs, ECGs and clinical laboratory parameters will be collected, tabulated, reviewed and recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers will be included in the study if they satisfy the following criteria:

* Healthy adult male or female volunteers (as determined by medical history, physical examination, laboratory test values, vital signs, an exercise stress test and electrocardiograms [ECGs] at screening) aged 18-45 years.
* Non-smokers from three months before receiving the first dose and for the duration of the study.
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Able and willing to receive rectal treatments.
* Able to voluntarily provide written informed consent to participate in the study.
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol.
* Female volunteers must be postmenopausal (for at least one year and confirmed by serum FSH at screening), surgically sterile, practising true sexual abstinence, or must use two highly effective methods of contraception as follows throughout the study until after post study physical examination: contraceptive implants, injectables, oral contraceptives, some intrauterine devices (IUDs), vasectomised partner and / or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository.
* Hormonal and IUD methods of contraception must be established for a period of 3 months prior to dosing and cannot be changed or altered during the study.
* Females of childbearing potential must have a negative pregnancy test at screening (β HCG) and at check-in.
* Sexually active male volunteers must use condoms with their partners throughout the study and for 90 days after completion of the study in addition to their partner's normal mode of contraception.
* Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
* The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study.

Exclusion Criteria:

Volunteers will be excluded if they fulfil any of the following criteria:

* Positive for HIV, hepatitis B, or hepatitis C as demonstrated by the results of testing at screening.
* History or presence of any significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
* History or presence of aortic stenosis or hypertrophic cardiomyopathy.
* History or presence of any clinically significant ano-rectal conditions as judged by the Investigator, clinically significant latex allergy or clinically significant drug allergy.
* Presence of any ECG abnormalities (during rest or during the exercise stress test).
* Pregnant or lactating females.
* Laboratory values at screening which are deemed to be clinically significant according to Bio-Kinetic Europe Ltd SOPs, unless agreed in advance by the Sponsor's Responsible Medical Officer and the Bio-Kinetic Investigator.
* Current or history of drug or alcohol abuse or a positive drugs of abuse test at screening or check in.
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Any significant illness during the screening period preceding entry into this study.
* Donation of blood or blood products within 90 days prior to study drug administration, or at any time during the study, except as required by this protocol.
* Strenuous exercise during study confinement and one week prior to dosing (with the exception of the screening exercise stress test).
* Consumption of alcoholic beverages within 24 hours of confinement. Abstinence is required during study confinement.
* Consumption of xanthine-containing products within 24 hours of confinement and during study confinement.
* Use of any disallowed concomitant medication, including over-the-counter items within 14 days prior to study drug administration until the end of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Steady state pharmacokinetics of NRL001 | 14 days

SECONDARY OUTCOMES:
Pharmacodynamic effects of NRL001 | 14 days
Safety will be assessed by recording adverse events (AEs), vital signs, 12-lead ECG, physical examinations and clinical laboratory tests. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, MRCGP MFPM, Principal Investigator — Bio-Kinetic Europe, Ltd.
Locations (1):
- Bio-Kinetic Europe Ltd, Belfast, United Kingdom

REFERENCES:
- [Derived] Bell D, Duffin A, Jacobs A, Pediconi C, Gruss HJ. A double-blind, placebo-controlled, randomised, parallel-group, dose-escalating, repeat dose study in healthy volunteers to evaluate the safety, tolerability, pharmacodynamic effects and pharmacokinetics of the once daily rectal application of NRL001 suppositories for 14 days. Colorectal Dis. 2014 Mar;16 Suppl 1:36-50. doi: 10.1111/codi.12544. PMID 24499495